CLINICAL TRIAL: NCT06706908
Title: Innovative Spinopelvic Solutions with Real-world Evidence
Acronym: INSPIRE
Status: Enrolling by invitation | Type: Observational
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 302022
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sacroiliac Joint Dysfunction; Sacroiliac Joint Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Health questionnaires — Participants are expected to complete a series of health questionnaires (i.e. numerical rating scale, Oswestry Disability Index) relevant to their treatment using a SI-BONE implant.

SUMMARY:
INSPIRE is a prospective decentralized study evaluating post-operative health outcomes in patients who undergo a procedure using implants manufactured by SI-BONE.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 at time of screening.
2. Patient will undergo a procedure utilizing an iFuse Implant family product.
3. Patient is comfortable communicating in written and spoken English.
4. Patient is willing and able to complete study questionnaires online, using either a smartphone, tablet, or computer.
5. Patient is willing and able to provide informed consent to participate

Exclusion Criteria:

1. Patient has fibromyalgia.
2. Patient has a pain pump.
3. Patient is currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an implant manufactured by SI-BONE.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported outcomes | From enrollment and at the following timepoints, 1-, 3-, 6-, and 12-months.
  Change in pain as rated on a numerical rating scale (NRS), 0 being no pain and 10 being the worst pain imaginable at baseline and follow-up timepoints.

SECONDARY OUTCOMES:
Change in patient reported outcomes | At the following timepoints: 1-, 3-, 6-, and 12-months.
  Change in patient satisfaction on a four point scale, with 0 being very dissatisfied and 3 being very satisfied at follow-up timepoints.

OTHER OUTCOMES:
Postoperative incidence of: | At the following timepoints, 1-, 3-, 6-, and 12-months.
  * Serious adverse events probably or definitely related to the implant of interest
  * Implant failures related to the implant of interest (e.g., revision surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Principal Investigator — SI-BONE
Locations (1):
- SI-BONE, Santa Clara, California, United States

IPD SHARING:
Plan to Share IPD: Undecided